CLINICAL TRIAL: NCT01114113
Title: Pilot Study: Assessment of Gastric and Intestinal Motility Following a Trigger Meal in Patients With Post Prandial Diarrhea
Brief Title: Assessment of Gastric Emptying Speed in Patients Who Experience Diarrhea Following a Trigger Meal
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of interest in participation by patients locally and lack of funding.
Sponsor: Money, Mary E., M.D. (Individual)
Responsible Party: Principal Investigator, Mary E. Money, M.D., Principal Investigator, Money, Mary E., M.D.
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2010IBS-G/D eval
Record Dates: First submitted 2010-04-25; First posted 2010-04-30 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Irritable Bowel Syndrome; Diarrhea
Keywords: IBS-D; Post meal Diarrhea; Trigger meals
MeSH Terms: conditions — Irritable Bowel Syndrome; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- non-trigger meal (Active Comparator): Measurement of intestinal transport eating a "non-trigger meal".
  Interventions: Device: SmartPill capsule
- "trigger meal baseline" (Active Comparator): Measurement of intestinal transport after eating a "trigger meal".
  Interventions: Device: SmartPill capsule
- "trigger meal" with placebo (Placebo Comparator): Measurement of intestinal transport with blinded placebo
  Interventions: Drug: pancelipase/placebo; Device: SmartPill capsule
- "trigger meal" with enzymes (blinded) (Active Comparator): Measurement of intestinal transport with blinded active enzyme capsule
  Interventions: Drug: pancelipase/placebo; Device: SmartPill capsule

INTERVENTIONS:
Drug: pancelipase/placebo — ZenPep 20000 units of lipase will be provided for the participant to take with a trigger meal or an identical placebo. This will only be given to those participants willing to consume 2 more identical "trigger meals" and will not be given for the initial baseline "non-trigger" and baseline "trigger meal". In both of these arms, patients will also be swallowing the SmartPill Capsule.
  Arms: "trigger meal" with enzymes (blinded); "trigger meal" with placebo
Device: SmartPill capsule — Measurement of a baseline, non-trigger meal intestinal transit by using the SmartPill capsule.
  Arms: non-trigger meal
Device: SmartPill capsule — Measurement of intestinal transit of a "trigger meal" baseline by using the SmartPill capsule
  Arms: "trigger meal baseline"
Device: SmartPill capsule — SmartPill capsule
  Arms: "trigger meal" with enzymes (blinded); "trigger meal" with placebo

SUMMARY:
The rapid diarrhea that patients experience who have diarrhea occurring after eating specific foods may be causing a "physiologic gastric dumping syndrome". This means that rather than the food being kept in the stomach for normal digestion, it rapidly goes into the small intestine and diarrhea occurs. This study is designed to measure how fast the food empties from the stomach when a person with this problem consumes a "regular diet", compared to a meal with a "triggering substance". Each participant will swallow a radio frequency capsule that with the different meals that will show how fast the food is traveling through the intestines in the different situations.

DETAILED DESCRIPTION:
Since some patients have found that pancreatic enzymes seem to ameliorate this diarrhea from occurring,willing participants will be asked to duplicate the "triggering meal" 2 more times. Once taking a pancreatic enzyme (active drug) with the meal and a second time taking an identical placebo. Neither the participant nor the study investigator will know which capsule is the active drug in this phase of the study. Willing participants will receive a small stipend each time they swallow the radio frequency capsule. This capsule is large, approximately twice the size of a vitamin pill so individuals must have no difficulties with swallow to participate nor any history of bowel obstruction or major surgery to the abdominal which might have caused adhesions.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have been diagnosed as having post prandial diarrhea for at least 5 years by his/her primary care physician or gastroenterologist and is believed to have no other medical condition that would cause this medical problem. Each person must be over 18 years old and have negative testing for Celiac Disease, a normal colonoscopy within 5 years of enrollment, and a normal Hgb and sedimentation rate within 6 months of enrollment in the trial.
2. The patient has provided documented written informed consent/authorization prior to initiation of any study-related procedure.
3. In addition, each patient must report experiencing the onset of urgent defecation within 1 hours of eating a specific trigger which is reproducible at least 90% of the time when consume.
4. The patient must be willing to comply with all of the study protocol.

Exclusion Criteria:

1. The patient has had any rectal bleeding or bloody stools within the last 2 years not completely evaluated by a physician. If rectal bleeding has occurred, and the patient wants to be considered for the study, the diagnostic workup must have clearly identified the etiology for the bleeding and excluded the medical conditions listed under 3 below. The patient must be willing to allow the Study team to obtain these records for verification of the diagnosis.
2. The patient has nocturnal bowel movements.
3. The patient has been diagnosed with or has a family history of any of the following: ulcerative colitis, Crohn's Disease, celiac disease, sprue, other inflammatory bowel disease or has a positive test for celiac disease on screening lab and has not had a full investigation performed to exclude celiac disease.
4. The patient has had unexplained anorexia or weight loss of more than 10% of body weight within 12 months of onset of study.
5. Prior GI surgery except of uncomplicated appendectomy and laparoscopic cholecystectomy or history of bowel obstruction or symptoms suggestive of such within the past 2 years.
6. The patient reports daily use of laxatives or stool softeners; use of fiber supplementation is permitted.
7. The patient is currently using pancrealipase. Previous use of pancrealipase in the past is allowed, but patients must be off either of the medication for at least 1 week or until the patient's symptoms of post prandial diarrhea returns before participating in the study.
8. Use of implanted or ambulatory electromechanical medical devices such as pacemakers, insulin pumps, and infusion pumps.
9. History of gastroparesis or chronic use of reglan.
10. Dysphagia to solid food and pills.
11. Previous gastro-esophageal surgery including vagotomy, fundoplication, gastric bypass or ulcer surgery.
12. Tobacco use within eight hours prior to capsule ingestion and during the 8 hour monitoring time.
13. Alcohol use within 24 hours prior to capsule ingestion and throughout the entire monitoring period (up to 72 hours).
14. BMI > 35
15. Female of childbearing age who is not practicing birth control and/or is pregnant or lactating. (Confirm with urine pregnancy test).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Duration of intestinal speed of a "trigger meal" compared to a non-trigger meal baseline. Optional study comparing intestinal speed of trigger meal using Pancrelipase compared to placebo. | 72 hour measurement per meal
  Data from the SmartPill radiofrequency capsule that is swallowed at the beginning of the different meals will be recorded and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Money, M.D., Principal Investigator — Washington County Hospital

REFERENCES:
- [Background] Money ME, Hofmann AF, Hagey LR, Walkowiak J, Talley NJ. Treatment of irritable bowel syndrome-diarrhea with pancrealipase or colesevelam and association with steatorrhea. Pancreas. 2009 Mar;38(2):232-3. doi: 10.1097/MPA.0b013e31817c1b36. No abstract available. PMID 19238028